CLINICAL TRIAL: NCT07057284
Title: DENtofacial TOxicity: Facilitating Advancement in Paediatric Cancer toxIcity Reporting And Liaison in Proton Beam Therapy. Stage 2 - Feasibility of Retrospective Toxicity Outcome Collection [DENTOFACIAL-PBT(2)]
Brief Title: DENTOFACIAL-PBT Stage 2 - Feasibility Study
Status: Enrolling by invitation | Type: Observational
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: The Christie NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: B02096
Record Dates: First submitted 2025-05-16; First posted 2025-07-09 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-06

CONDITIONS: Head and Neck Cancer; Radiotherapy Side Effect; Adverse Effect of Radiation Therapy; Childhood Cancer; Dental Developmental Disorders and Anomalies; Facial Deformity; Jaw; Developmental Disorder; Radiation Toxicity
MeSH Terms: conditions — Head and Neck Neoplasms; Radiation Injuries; Neoplasms; Congenital Abnormalities; Developmental Disabilities | interventions — Radiography, Panoramic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Orthopantomogram (or a set of Lateral Oblique Radiographs) — A dental assessment will be conducted on eligible participants who still attend annual review appointments in the Oncology Departments at the Royal Manchester Children's Hospital or at The Christie NHS Foundation Trust (approximately 10% of eligible study population). The dental assessment will include the following: a tooth chart, a basic periodontal examination (BPE), a brief orthodontic assessment (incisor, molar and skeletal classification including any asymmetry), caries assessment and an assessment of any dental development disturbances. Clinical photographs of the teeth and face will be taken with a patient's consent. If clinically justified, an OPT will be taken. If cooperation for an OPT proves challenging, lateral obliques as an alternative radiographic image modality will be considered.

SUMMARY:
What is the health problem? Proton beam therapy (PBT), a type of radiotherapy treatment, can be especially beneficial to children and teenagers with cancer. PBT works by damaging cancer cells, but it can also damage healthy parts of the body nearby. This can include the teeth and jaws if the cancer is in the head and neck region. Unfortunately, the investigators do not yet fully understand the potential side effects of PBT on the teeth or jaws.

What is the aim? The DENTOFACIAL-PBT research project aims to learn about the side effects to the teeth and jaws in children treated with PBT. This stage of the research aims to determine how frequently issues ('toxicities') in the development of the teeth and growth of the jaws have occurred in previously treated patients. DENTOFACIAL-PBT is funded by the National Institute for Health and Care Research.

How is the researched being approached? The investigators will ask head and neck childhood cancer survivors treated with PBT overseas or in Manchester to support this research. Surveys will be sent initially, asking questions about their teeth and jaws after treatment. If interested, these survivors can be involved in the next part of this stage, which is a mixed-methods feasibility study. This will involve online interviews and dental assessments with some and the collection of dental information from a participant's dentist. Radiation dose to the teeth and the jaw bones will then be linked to any side effects seen.

What will be the outcome? The information gained in this study will allow the research team to look at how age, location and amount of dose given affects the toxicities seen. Information learnt will help develop the final stage of the DENTOFACIAL-PBT study. In this, a new toxicity reporting tool will be developed which aims to improve the communication between dentists, doctors, and cancer patients.

DETAILED DESCRIPTION:
The overall aim is to ascertain if it is feasible to determine the prevalence of adverse effects to the teeth and jaws in the United Kingdom National Health Service cohort of childhood head and neck cancer survivors treated with proton beam therapy using a mixed methods study. This will involve data being collected both retrospectively and prospectively. This study is being hosted by Manchester University NHS Foundation Trust with the support of the Proton Clinical Outcomes Unit at The Christie NHS Foundation Trust.

RESEARCH QUESTIONS:

[RQ-1]: How often have adverse effects to the teeth and jaws occurred in UK childhood head and neck cancer patients treated with proton beam therapy at The Christie NHS Foundation Trust and overseas in the NHS Proton Overseas Programme? [RQ-2] Is it practical to collect data on side effects to the teeth and jaws in this group of patients? [RQ-3] Is it possible to reliably contour the maxilla, mandible and the teeth on treatment planning computed tomography images to extract the radiation dose to these structures? [RQ-4] How should dental outcomes in childhood head and neck cancer patients treated with proton beam therapy be monitored? [RQ-5] Is it possible to link side effects reported by patients to their treatment dose? [RQ-6] Do side effects reported by patients align with those reported by their dentist? [RQ-7] What is the effect of age at the time of treatment on dentofacial development? [RQ-8] What is the effect of radiation dose on dentofacial development? [RQ-9] Is the QoL in childhood head and neck cancer survivors different in those with and without reported / identified dentofacial toxicities?

STUDY DESIGN:

A mixed methods, cross-sectional, self-administered survey has been developed. This is to be completed once by an eligible study participant. The survey contains pre- and post-treatment questions focused on the teeth and jaws, as well as including select scales from the FACE-Q™ Craniofacial module to collect HRQoL data. Participants aged 16 years or older will be directed to complete the survey individually. For participants aged less than 16 years old at the time of survey distribution, an individual with parental responsibility will be directed to complete the survey alongside their child. At the end of the survey, participants will be asked if they would be interested in being involved in a feasibility study regardless of whether they have reported a dentofacial toxicity. If a survey respondent enrols in the feasibility study, their completed survey will be linked to the data collected in the feasibility study. If a survey respondent does not enrol in the feasibility study, no patient-identifiable data will be collected, therefore their survey answers will be anonymous.

This feasibility study will aim to retrospectively analyse paediatric HNC patients treated with PBT to determine the prevalence of dentofacial toxicities, the feasibility of correlating PROs to PBT dosimetric data to establish dose-effect relationships, and to determine if it is possible to compare PROs to those reported by dental professionals. Information on the development of a participant's teeth and jaws will be requested from their dentist (if applicable). Further insight into the beliefs and concerns of patients will be elicited through virtual semi-structured qualitative interviews, which will adopt a 'palette of methods' approach. Additionally, individuals residing in the Greater Manchester area who attend an annual review with an Oncologist will be offered the opportunity to have a dental assessment at their next scheduled visit (n = approximately 25 patients). This will not only provide an additional opportunity for study recruitment should an individual not already be enrolled, but it will allow additional data collection on dental outcomes in this cohort. There will be no randomisation, blinding or masking of recruited participants.

Once a participant has consented and is enrolled into the study, the research team will conduct the following steps:

(A) Notify the Proton Clinical Outcomes Unit of a participant's enrolment and request patient identifiable treatment planning data from the clinical system at The Christie. For example, this data will include, sex, age at treatment, diagnosis, subsite, treatment location, chemotherapy history, surgery history and follow-up time. This will include any data collected on select AEs/toxicities, specifically 'musculoskeletal deformity', 'dental development disorders', 'dental caries' and 'periodontal disease' as graded in the 'Common Terminology Criteria for Adverse Effects' (CTCAE) version 5.0 (2017).

(B) Details of the participant's dentist (if registered) will be requested directly from the participant at the start of the study. Once these details are available, a letter will be sent to a participant's dentist outlining the following about the study: its aims, source of funding, ethical approval status, information requests, timeframes, and plans for dissemination of findings. Only information on the development of the teeth and jaws will be requested. This will include requesting relevant radiographs (X-Rays) that show the patient's teeth before (if available) and after treatment.

(C) Assessment of dental radiographs and dental clinical photographs (if available) from the clinical system at The Christie or MFT.

(D) Qualitative Interviews on MS Teams: Further insight into CCS thoughts and experiences will be elicited through virtual semi-structured interviews with a purposeful sample of participants to enhance and enrich the quantitative data.To enable participants with a variety of different skill sets and confidence levels to participate, the researcher will offer a list of methods for the individual to opt into. It is recognised that children are key stakeholders in this study and that their perspectives on dentofacial toxicities need to be considered. Allowing alternative approaches to participation to a traditional one-to-one interview may empower participants, thus making the research more inclusive.

Participation in the interviews could occur in five ways:

1. Individual participation of a CCS now aged 16 years or older,
2. A CCS now aged 16 years or older alongside a friend or family member for moral support.
3. Individual participation of a person with parental responsibility for an eligible participant aged less than16 years,
4. Participation of a person with parental responsibility alongside an eligible participant aged less than 16 years.
5. Participation of a person with parental responsibility alongside a friend or family member for moral support (without CCS) [healthy volunteer/s].

(E) Dental assessment and collection of PROMs data on established Oncology clinics: 10% (n = approximately 25) of the eligible study cohort attend a follow-up clinic in Manchester to review any late treatment adverse effects once a year. These established clinics are held at The Royal Manchester Children's Hospital (RMCH) [for individuals <16 years old, known to patients as a "follow-up clinic"] and at The Christie NHS Foundation Trust [for individuals >16 years old, known to patients as a "late effects clinic"]. Prior to contacting eligible participants, the radiation plan will be checked to confirm that radiation dose to the maxilla, mandible and/or teeth was received. If radiation was not delivered to these structures, a participant will not be contacted. Eligible participants attending these clinics will be contacted with a separate PIS, outlining the opportunity to see a dentist at their next scheduled clinical visit and to have a dental assessment, which will include an orthopantomogram (OPT).

ELIGIBILITY:
INCLUSION CRITERIA FOR THE SURVEY AND FEASIBILITY STUDY (steps A-D):

* (i) CCS previously diagnosed with HNC. This includes the oral cavity (lips, front two-thirds of the tongue, the gums, the lining inside the cheeks and lips, the floor of the mouth, under the tongue and the hard palate), the throat (nasopharynx, oropharynx and hypopharynx), the voice box (larynx), the paranasal sinuses, nasal cavity and the salivary glands
* (ii) Any sex.
* (iii) Currently a minimum age of 2 years.
* (iv) Treated with PBT at The Christie PBT centre (Manchester, UK) or treated overseas with PBT as part of the NHS Proton Overseas Programme.
* (v) Completed treatment with PBT when aged 15 years and under.
* (vi) Completed treatment with PBT more than 12 months ago.
* (vii) Able and willing to provide informed consent or informed consent provided by a parent or person with parental responsibility in law for a child currently aged less than 16 years old who meets the inclusion criteria outlined in (i) to (vi).
* (viii) Language - Capacity to translate study documents and conduct interviews in the following languages: English, Arabic, Chinese, Dutch, French, German, Italian, Portuguese, Russian, Spanish and Turkish.

INCLUSION CRITERIA FOR STEP E OF THE FEASIBILITY STUDY

* (i) CCS previously diagnosed with HNC. This includes the oral cavity (lips, front two-thirds of the tongue, the gums, the lining inside the cheeks and lips, the floor of the mouth, under the tongue and the hard palate), the throat (nasopharynx, oropharynx and hypopharynx), the voice box (larynx), the paranasal sinuses, nasal cavity and the salivary glands.
* (ii) Any sex.
* (iii) Currently a minimum age of 2 years old for a clinical assessment without a radiograph to be conducted. The minimum age of a participant that a radiograph will be attempted at is 3 years old.
* (iv) Referred for PBT treatment by the Oncology team at The Royal Manchester Children's Hospital.
* (v)Treated with PBT at The Christie PBT centre (Manchester, UK) or treated overseas with PBT as part of the NHS Proton Overseas Programme.
* (vi) Completed treatment with PBT when aged 15 years and under.
* (vii) Completed treatment with PBT more than 12 months ago.
* (viii) Attending annual review clinics at either The Royal Manchester Children's Hospital ("follow-up clinic") or at The Christie NHS Foundation Trust ("late effects clinic") with the Oncology team.
* (ix) Able and willing to provide informed consent or informed consent provided by a parent or person with parental responsibility in law for a child currently aged less than 16 years old who meets the inclusion criteria outlined in (i) to (viii).
* (x) Language - English, Arabic, Chinese, Dutch, French, German, Italian, Portuguese, Russian, Spanish and Turkish.

EXCLUSION CRITERIA FOR THE SURVEY AND FEASIBILITY STUDY (steps A-D)

* (i) Deceased patients
* (ii) Aged greater than or equal to 16 years old at the time of diagnosis
* (iii) Currently aged less than 2 years old
* (iv) Completed PBT less than 12 months ago. (Although the minimal follow-up time for dentofacial toxicities to develop is unknown, it is felt that setting this restriction will enable eligible participants to have processed their treatment and had multiple reviews within this first year. This criterion of follow-up was discussed with the developed patient advisory group and this timeframe was felt to be the most appropriate).
* (v) Individuals treated with PBT overseas but not referred from a UK centre (not in the Proton Overseas Programme). For example, individuals whose care was privately funded or funded by an insurance company. The PCO Database maintained by the PCOU will not hold outcome data for privately funded patients.
* (vi) A parent or person with parental responsibility in law for a CCS now aged greater than 16 years old.
* (vii) Exclusion of any participant who does not speak a language specified in the inclusion criteria.

EXCLUSION CRITERIA FOR STEP E OF THE FEASIBILITY STUDY

* (i) Deceased patients
* (ii) Aged greater than or equal to 16 years old at the time of diagnosis
* (iii) Currently aged less than 2 years old
* (iv) Completed PBT less than 12 months ago.
* (v) Individuals treated with PBT overseas but not referred from a UK centre (not in the Proton Overseas Programme). For example, individuals whose care was privately funded or funded by an insurance company.
* (vi) No radiation delivered to the maxilla, mandible and/or teeth.
* (vii) A parent or person with parental responsibility in law for a CCS now aged greater than 16 years old.
* (viii) Living outside of the Greater Manchester region and not attending routine annual clinics with the Oncology team at The Royal Manchester Children's Hospital or at The Christie NHS Foundation Trust.
* (ix) Exclusion of any participant who does not speak a language specified in the inclusion criteria.

Ages: 2 Years to 32 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Childhood head and neck cancer survivors who were treated with proton beam therapy either in the National Health Service Proton Overseas Programme or at The Christie NHS Foundation Trust.
Sampling Method: Non-Probability Sample
Enrollment: 255 (Estimated)
Dates: Start 2026-01-16 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate and number of participants with complete datasets. | From enrolment until study completion, an average of 1 year.
  Usability and completeness of the study data. A 'complete dataset' for a participant refers to the following: completed survey, cancer diagnosis, treatment and follow-up information, pre- and post- radiotherapy dental radiographs, dental information from a participants dentist and extracted dentofacial dosimetric statistics.
Presence of dentofacial toxicities | Through study completion, an average of 1 year.
  Prevalence of dentofacial toxicities in the UK cohort of paediatric HNC patients treated with PBT.

SECONDARY OUTCOMES:
Patient perspectives on dentofacial development and toxicities. | From enrolment to the completion of the last study interview, an average of 1 year.
  Generation of themes during the analysis of qualitative interviews.
Dental health seeking behaviour and practices. | From enrolment to the completion of the last study interview, an average of 1 year.
  Generation of themes via qualitative interviews.
Patient-reported dentofacial toxicity outcomes. | From enrolment to study completion, an average of 1 year.
  Dose-effect relationship determination from PROs and PBT dosimetric data. Correlation of clinician-reported outcomes to patient-reported outcomes.
Clinician-reported dentofacial toxicity outcomes | From enrolment to study completion, an average of 1 year.
  Dose-effect relationship determination from PROs and PBT dosimetric data. Correlation of clinician-reported outcomes to patient-reported outcomes.
Extracted radiation dose statistics. | Following collection of all data (30/09/2026)
  and PBT dosimetric data. Correlation of clinician-reported outcomes to patient-reported outcomes.
Dentofacial development and age | Following collection of all data (30/09/2026).
  The effect of chronological age at treatment on dentofacial development.
Dentofacial development and radiation dose. | Following completion of all data (30/09/2026).
  The effect of mean radiation dose on dentofacial development.
Health-related quality of life (HRQoL) assessed using scales from the FACE-Q™ Craniofacial module. | Through study completion, an average of 1 year.
  HRQoL outcomes reported via the FACE-Q Craniofacial Module (unabbreviated title). Ten scales from this module will be used, specifically, 'face', 'jaws', 'smile', 'teeth', 'cheeks', 'nose', 'facial', 'appear distress', 'social' and 'psychological'. There is no overall or total FACE-Q score. The FACE-Q is composed of independently functioning scales, checklists, and stand-alone items. To score a scale, raw scores for the set of items in a scale are added together to produce a total raw score. A conversion table will then be used to convert the total raw score into a score that ranges from 0 (worst) to 100 (best). Higher scores reflect a better outcome.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Manchester University NHS Foundation Trust, Manchester
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No